CLINICAL TRIAL: NCT01261676
Title: Current Dutch Practice on Caesarean Sections: Identification of Barriers and Facilitators for Optimal Care.
Acronym: SIMPLE
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 09-4-047; 17100.3006 (Other Grant/Funding Number: zonMW)
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2012-10-30 (Estimated); Status verified 2012-10

CONDITIONS: Caesarean Section
Keywords: caesarean section; labour, obstetric; implementation guidelines; quality indicators

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Caesarean section
  Interventions: Other: Implementation aids
- Vaginal birth (control)
  Interventions: Other: Implementation aids

INTERVENTIONS:
Other: Implementation aids — An implementation strategy to improve outcome for women in labour will be developed depending on the outcome of the current care study and the barrier and facilitator analysis.The strategy will be executed and evaluated in a controlled before-and-after study in 12 hospitals (6 intervention, 6 control)

SUMMARY:
Caesarean (CS) delivery rates in the Netherlands increased from 5 to 15% the last 20 years. CSs have no clear benefit for overall neonatal outcome and are associated with higher maternal complications and high costs. Dutch guidelines offer clear recommendations on factors that have a direct effect on the decision to perform a CS.

Hypothesis: there is incomplete adherence to the recommendations from the guidelines on CS among Dutch gynaecologists.

This study consists of four phases:

1. Development of quality indicators: A set of quality indicators regarding the process, structure and outcome of care will be developed according to the RAND-modified Delphi method. A representative, national expert panel consisting of 12 to 15 obstetricians and midwives will participate.
2. Current care study: The current Dutch care will be studied in 20 hospitals (N=80 gynaecologists). 1000 files on performed CSs are analyzed regarding the adherence to the developed quality indicators. To get insight into Dutch practices compared to international data, basic obstetrical data will be extracted from the delivery database.
3. Barrier analysis: A barrier analysis will be carried out based on the results of the current care study. Two groups of hospitals will be identified in the upper and lower extremes of the 'adherence distribution': 5 hospitals with the lowest and 5 hospitals with the highest adherence scores. Factors that determine the decision to perform a CS or not (barriers and facilitators) will be analyzed in both groups using semi-structured interviews among 15-20 professionals and 15-20 patients. A questionnaire will be used to study the 'prevalence' of these factors among all obstetric gynaecologists in the Netherlands and among 200 patients.
4. Controlled before- and-after (CBA) study: Based on the outcomes of the current care study and the barrier analysis, a tailor made implementation strategy will be developed in order to increase adherence to the CS quality indicators. Target groups will be selected with focus on women with both a high incidence of the indicator and low indicator adherence. The strategy will be executed and evaluated in a CBA-study in 12 hospitals (6 intervention, 6 control) in terms of effectiveness, experiences and costs. The sample size will be dependent on the target group and adherence to the quality indicators regarding this target group. These data will be available after performing the current care and the barrier study.

ELIGIBILITY:
Inclusion Criteria:

* A previous caesarean section in a 3-4 month time period.

Exclusion Criteria:

* Major congenital malformality
* Fetal death prior to onset of delivery
* Duration of pregnancy less than 24 weeks of gestation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Development of quality indicators: 12-15 obstetricians and midwives
  2. Current care study: All women (1000) who underwent a CS in one of the 20 participating hospitals during the study period (3-4 months). All hospitals participate in the Dutch consortium and consist of university teaching-, non-university teaching- and non-university-non-teaching hospitals.
  3. Barrier analysis: Qualitative: 15-20 professionals and 15-20 patients from the hospitals in the upper and lower extremes of the 'adherence distribution'. Quantitative: obstetricians in the Netherlands and 200 experienced patients.
  4. CBA study: depending on the outcome of phase 2 and 3 of the study, the implementation strategy will be designed for a target group with low guideline adherence and high incidence.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-12; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
1) Development of quality indicators: development of a valid set of quality indicators for measuring current Dutch care on caesarean sections | December 2010 - October 2013
2) Current care study: The main outcome is the adherence to the quality indicators regarding the process, structure and outcome (maternal and fetal) of care | December 2010 - October 2013
3) Barrier and facilitator analysis: Identification of barriers and facilitators to perform a caesarean section | December 2010 - October 2013
4) Controlled before-and-after study: effectiveness of the implementation strategy defined as observed increase in adherence between the intervention and control hospitals and actual CS rates in both groups | December 2010 - October 2013

SECONDARY OUTCOMES:
1) Development of quality indicators: no secondary outcomes | December 2010 - October 2013
2) Current care study: International comparison | December 2010- October 2013
  Dutch practice as compared to international data (Robson criteria)
3) Barrier and facilitator analysis: no secondary outcomes | December 2010-October 2013
4) Controlled before-and-after study: experiences and satisfaction of health care providers and patients with the implementation strategy and applicability and costs of the strategy | December 2010-October 2013

CONTACTS AND LOCATIONS:
Overall Officials: Hubertina CJ Scheepers, Ph.D., Principal Investigator — Maastricht University Medical Center
Locations (20):
- Netherlands (20):
  - Ziekenhuisgroep Twente, Almelo
  - Flevo Ziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Academisch Medisch Centrum, Amsterdam
  - Gelreziekenhuizen, Apeldoorn
  - Rijnstate Ziekenhuis, Arnhem
  - Ijsselland Ziekenhuis, Capelle Aan Den Ijjsel
  - Catharina-ziekenhuis, Eindhoven
  - University Medical Centre Groningen, Groningen
  - Röpcke-Zweers Ziekenhuis, Hardenberg
  - Atrium Medisch Centrum Parkstad, Heerlen
  - Elkerliek Ziekenhuis, Helmond
  - Tergooiziekenhuizen, Hilversum
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Universitair Medisch Centrum St. Radboud, Nijmegen
  - Orbis Medisch Centrum, Sittard
  - Universitair Medisch Centrum Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - Sint Jansgasthuis, Weert
  - Zaans Medisch Centrum, Zaandam

REFERENCES:
- [Derived] Melman S, Schoorel EN, Dirksen C, Kwee A, Smits L, de Boer F, Jonkers M, Woiski MD, Mol BW, Doornbos JP, Visser H, Huisjes AJ, Porath MM, Delemarre FM, Kuppens SM, Aardenburg R, Van Dooren IM, Vrouenraets FP, Lim FT, Kleiverda G, van der Salm PC, de Boer K, Sikkema MJ, Nijhuis JG, Hermens RP, Scheepers HC. SIMPLE: implementation of recommendations from international evidence-based guidelines on caesarean sections in the Netherlands. Protocol for a controlled before and after study. Implement Sci. 2013 Jan 3;8:3. doi: 10.1186/1748-5908-8-3. PMID 23281646